CLINICAL TRIAL: NCT00474240
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Safety and Efficacy of the Combination of AEGR-733 (Formerly BMS201038) and Atorvastatin 20 mg vs. Monotherapy in Subjects With Moderate Hypercholesterolemia
Brief Title: AEGR-733 and Atorvastatin 20 mg vs. Monotherapy in Moderate Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEGR-733-003
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2013-01

CONDITIONS: Hypercholesterolemia
Keywords: cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin; BMS201038

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: Atorvastatin 20 mg
- 3 (Experimental)
  Interventions: Drug: AEGR-733 5 mg
- 4 (Experimental)
  Interventions: Drug: AEGR-733 10 mg
- 5 (Experimental)
  Interventions: Drug: AEGR-733 5 mg + atorvastatin 20 mg
- 6 (Experimental)
  Interventions: Drug: AEGR-733 10 mg + atorvastatin 20 mg

INTERVENTIONS:
Drug: Atorvastatin 20 mg
  Arms: 2
Drug: AEGR-733 5 mg
  Arms: 3
Drug: AEGR-733 10 mg
  Arms: 4
Drug: Placebo
  Arms: 1
Drug: AEGR-733 5 mg + atorvastatin 20 mg
  Arms: 5
Drug: AEGR-733 10 mg + atorvastatin 20 mg
  Arms: 6

SUMMARY:
The purpose of this study is to test the effectiveness of the study drug, AEGR-733 alone and in combination with the medication, atorvastatin (Lipitor), on cholesterol in volunteers with moderately high cholesterol.

DETAILED DESCRIPTION:
Recent studies suggest more intensive cholesterol lowering treatment for people at very high risk of a heart attack, specifically for patients who have heart disease plus major risk factors. Available medications used alone at even the highest approved doses are not expected to reach these new target recommendations for cholesterol in a large number of subjects. Thus, the development of new medications that can provide additional cholesterol lowering may be beneficial.

This study tests the effectiveness of different doses of the study drug, AEGR-733 alone and in combination with the approved cholesterol lowering drug, atorvastatin (Lipitor), on cholesterol. Volunteers will be randomized to one of 6 different study treatments and will take the assigned medication (3 capsules daily) for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 70 years.
2. Elevated LDL cholesterol based on risk factors for cardiovascular disease or presence of cardiovascular disease

Exclusion Criteria:

1. Women who are pregnant, lactating, planning to become pregnant, or women of childbearing potential who have not successfully been using acceptable contraceptive methods over the previous 3 months, e.g., intrauterine device (IUD) and barrier method plus spermicide.
2. Uncontrolled hypertension
3. History of chronic kidney problems
4. History of liver disease
5. Positive for Hepatitis B or Hepatitis C.
6. Any major surgical procedure occurring less than 3 months ago
7. Cardiac insufficiency
8. History of a malignant cancer (other than basal cell or squamous cell carcinoma of the skin that has been removed) within the previous 5 years.
9. Regular alcohol use >1 drink per day.
10. Regular consumers of grapefruit juice, or currently taking the following medications: cyclosporine, itraconazole, ketoconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, and nefazodone.
11. Use of other cholesterol lowering medications that cannot be stopped.
12. Heart attack or stroke within the previous 6 months
13. Diabetes Mellitus
14. Body mass index (BMI) ≥ 40 kg/m2.
15. Significant gastrointestinal symptoms, such as irritable bowel syndrome.
16. Current use of fish oils, niacin, and herbal weight loss products that cannot be stopped.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Jacksonville Center for Clinical research, Jacksonville, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Renstar Medical Research, Ocala, Florida
  - North Georgia Clinical Research, Woodstock, Georgia
  - Radiant Research, Chicago, Illinois
  - Medsphere Medical Research Center, Evansville, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Maine Research Associates, Auburn, Maine
  - Health Trends Research, Baltimore, Maryland
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Sterling Research Group, Cincinnati, Ohio
  - Coastal Carolina Research Center, Goose Creek, South Carolina
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Diabetes and Glandular Disease Research, Dallas, Texas
  - Hampton Roads Center for Clinical Research, Norfolk, Virginia
  - National Clinical Research, Richmond, Virginia

REFERENCES:
- [Background] Cuchel M, Bloedon LT, Szapary PO, Kolansky DM, Wolfe ML, Sarkis A, Millar JS, Ikewaki K, Siegelman ES, Gregg RE, Rader DJ. Inhibition of microsomal triglyceride transfer protein in familial hypercholesterolemia. N Engl J Med. 2007 Jan 11;356(2):148-56. doi: 10.1056/NEJMoa061189. PMID 17215532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed from 05 November 2007 to 04 August 2008 at 17 medical clinics within the United States.
Pre-assignment Details: Subjects who were previously on a lipid lowering therapy underwent a 5-week washout period. All subjects were on a low-fat diet (<30% calories from fat) starting 5 weeks prior to study drug treatment and continuing for the duration of the study.
Groups:
- Placebo: Placebo capsule taken orally once daily
- Atorvastatin 20 mg: Atorvastatin 20 mg taken orally once daily
- AEGR-733 5 mg: AEGR-733 5 mg taken orally once daily
- AEGR-733 10 mg: AEGR-733 10 mg taken orally once daily
- AEGR-733 5 mg + Atorvastatin 20 mg: One capsule of AEGR-733 5 mg and 1 capsule of Atorvastatin 20 mg taken orally once daily
- AEGR-733 10 mg + Atorvastatin 20 mg: One capsule of AEGR-733 10 mg and 1 capsule of Atorvastatin 20 mg taken orally once daily
Period: Overall Study
Arm/Group | Placebo | Atorvastatin 20 mg | AEGR-733 5 mg | AEGR-733 10 mg | AEGR-733 5 mg + Atorvastatin 20 mg | AEGR-733 10 mg + Atorvastatin 20 mg
Started | 27 | 26 | 26 | 26 | 26 | 26
Completed | 26 | 25 | 17 | 10 | 18 | 8
Not Completed | 1 | 1 | 9 | 16 | 8 | 18
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 9 | 14 | 5 | 16
Not completed — Removed due to lab value | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atorvastatin 20 mg | AEGR-733 5 mg | AEGR-733 10 mg | AEGR-733 5 mg + Atorvastatin 20 mg | AEGR-733 10 mg + Atorvastatin 20 mg | Total
Number analyzed (Participants) | 27 | 26 | 26 | 26 | 26 | 26 | 157
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53 (11.1) | 56 (8.4) | 56 (8.3) | 54 (11.6) | 51 (10.1) | 53 (9.7) | 54 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 16 | 16 | 10 | 16 | 87
  Male | 14 | 10 | 10 | 10 | 16 | 10 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 3 | 3 | 0 | 7
  Not Hispanic or Latino | 27 | 26 | 25 | 23 | 23 | 26 | 150
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 2 | 4 | 5 | 3 | 23
  White | 22 | 21 | 23 | 21 | 18 | 22 | 127
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 3 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 26 | 26 | 26 | 26 | 157

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at 8 Weeks
Time Frame: Atfer 8 weeks on study drug
Population: Intent To Treat
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Atorvastatin 20 mg | AEGR-733 5 mg | AEGR-733 10 mg | AEGR-733 5 mg + Atorvastatin 20 mg | AEGR-733 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 25 | 24 | 18 | 10 | 18 | 9
Percent Change | 2 (11.2) | -42 (16.4) | -16 (17.3) | -37 (23.0) | -47 (19.2) | -50 (28.0)

2. Secondary Outcome: Percent Change From Baseline of Other Lipids
Time Frame: After 8 weeks of study drug
Population: Intent To Treat
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Atorvastatin 20 mg | AEGR-733 5 mg | AEGR-733 10 mg | AEGR-733 5 mg + Atorvastatin 20 mg | AEGR-733 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 26 | 25 | 19 | 10 | 18 | 9
Percent
  Percent change from baseline in total cholesterol | 2 (9.9) | -30 (12.4) | -18 (14.6) | -33 (19.0) | -37 (15.3) | -40 (20.7)
  Percent change from baseline in total Apo B | 0 (11.0) | -34 (13.0) | -17 (12.4) | -36 (21.9) | -41 (16.9) | -46 (19.8)
  Percent change from baseline in non-HDL-C | 2 (10.3) | -38 (15.8) | -19 (17.1) | -36 (26.0) | -45 (17.7) | -48 (24.5)

ADVERSE EVENTS:
Arm/Group | Placebo | Atorvastatin 20 mg | AEGR-733 5 mg | AEGR-733 10 mg | AEGR-733 5 mg + Atorvastatin 20 mg | AEGR-733 10 mg + Atorvastatin 20 mg
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 1/26 | 1/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 17/27 | 15/26 | 23/26 | 23/26 | 21/26 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Atorvastatin 20 mg (N=26) | AEGR-733 5 mg (N=26) | AEGR-733 10 mg (N=26) | AEGR-733 5 mg + Atorvastatin 20 mg (N=26) | AEGR-733 10 mg + Atorvastatin 20 mg (N=26)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Atorvastatin 20 mg (N=26) | AEGR-733 5 mg (N=26) | AEGR-733 10 mg (N=26) | AEGR-733 5 mg + Atorvastatin 20 mg (N=26) | AEGR-733 10 mg + Atorvastatin 20 mg (N=26)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 16 (16) | 15 (15) | 11 (11) | 20 (20)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (5) | 7 (7) | 5 (5) | 14 (14)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 4 (4)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Nasopharyngitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatice Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthenia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood Urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastric Dilatation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Potassium Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study AEGR-733-003, initiated in May 2007, was halted, and restarted under an amended Protocol in November 2007.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Information is unavailable.